CLINICAL TRIAL: NCT03029650
Title: Absolute Bioavailability/Pharmacokinetic and Residual Drug Analysis of the Transderm Scōp System in Healthy Adults
Brief Title: Scopolamine Patch Pharmacokinetics in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Nicole K Brogden, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 201506778
Record Dates: First submitted 2017-01-17; First posted 2017-01-24 (Estimated); Results first posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Healthy
Keywords: Peer Review; Research
MeSH Terms: interventions — Scopolamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transderm Scop® (Active Comparator): Each of the subjects will receive a single intravenous dose of 0.4 mg scopolamine hydrobromide and will wear the Transderm Scop® patch (1.5 mg) for 3 days in a crossover design with adequate washout in between. Subjects will be randomized to Group 1 (Transderm Scop® first followed by intravenous scopolamine hydrobromide) and remaining subjects will be randomized to Group 2 (intravenous scopolamine hydrobromide first followed by Transderm Scop®).
  Interventions: Drug: Transderm Scop®; Drug: Intravenous scopolamine hydrobromide
- Intravenous scopolamine hydrobromide (Experimental): Each of the subjects will receive a single intravenous dose of 0.4 mg scopolamine hydrobromide and will wear the Transderm Scop® patch (1.5 mg) for 3 days in a crossover design with adequate washout in between. Subjects will be randomized to Group 1 (Transderm Scop® first followed by intravenous scopolamine hydrobromide) and remaining subjects will be randomized to Group 2 (intravenous scopolamine hydrobromide first followed by Transderm Scop®).
  Interventions: Drug: Transderm Scop®; Drug: Intravenous scopolamine hydrobromide

INTERVENTIONS:
Drug: Transderm Scop® — TDDS dosage is 1.5 mg/72 hrs
Drug: Intravenous scopolamine hydrobromide — 0.4 mg via intravenous injection

SUMMARY:
The study to be performed will utilize already FDA-approved marketed products in healthy adults for the purpose to generate data for establishing rate of drug delivery of Transderm Scop® TDDS (transdermal drug delivery system) in healthy adults and to ensure safety of individuals utilizing these types of products.

DETAILED DESCRIPTION:
Transdermal drug delivery systems (TDDS) available in the form of patches are convenient, attractive, and easy to use systems. Scopolamine patches are very popular TDDS available on the United States market today. Accurate determination of the rate and extent of drug release and absorption is crucial to ensure the safety of individuals using these and other types of patches. Delivery rate can be determined early in the development process by using in vitro skin flux permeation studies, and later in humans by accurately quantifying residual drug from patches post-wear and in pharmacokinetic studies. In this proposal, the investigators will employ two types of evaluation to determine the rate and extent of drug release and absorption from RLD (reference listed drug) Transderm Scop® TDDS (transdermal drug delivery system), namely residual drug analysis post-wear and pharmacokinetic analysis in healthy adult volunteers. In addition, the investigators will compare the plasma drug concentrations following patch and intravenous administration of Scopolamine, in order to determine the absolute bioavailability of these patches. The investigators will conduct residual drug analysis of TDDS following in vivo wear using highly sensitive validated quantification methods. Positive outcomes of this project will identify appropriate methods to determine the rate and extent of drug release and absorption from TDDS, and will help regulatory agencies in the development of Guidances for Industry regarding the characterization of drug release and absorption kinetics to ensure the safety of individuals utilizing these types of products

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant women of any ethnic background between the age of 18 and 65 years old.
2. Subjects must be non-smokers (must have refrained from the use of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, gum, patch or electronic cigarettes) over the previous 12 months and are not currently using tobacco products.
3. Provide written informed consent before initiation of any study procedures.
4. Available for follow-up for the planned duration of the study.
5. Able to communicate well with the investigators.
6. Able to adhere to the study protocol schedule, study restrictions and examination schedule.
7. Subjects who are within their ideal body weight (BMI between 18-29.9 kg/m2).
8. Demonstrate comprehension of the protocol procedures and knowledge of study, as demonstrated a study member filling out a consent checklist form to verify that the subject understands all aspects of the study including the purpose, procedures, risks and benefits.
9. Subjects deemed to be healthy as judged by the Medically Accountable Investigator (MAI) and determined by medical history, physical examination, and medication history.
10. Negative urine drug screening test.
11. Have a normal blood pressure (systolic: 90-140 mmHg; diastolic: 50-90 mmHg) and heart rate (55-100 bpm).
12. Have normal screening laboratories for WBC, Hgb, Hct, platelets, sodium, potassium, chloride, bicarbonate, BUN, creatinine, ALT, AST, and total bilirubin.
13. Have normal screening laboratories for urine protein and urine glucose.
14. Female subjects must be of non-childbearing potential (defined as surgically sterile [i.e. history of hysterectomy or tubal ligation] or postmenopausal for more than 1 year [no bleeding for 12 consecutive months]), or if of childbearing potential must be non-pregnant at the time of enrollment and on the morning of the first day of each study treatment session, and must agree to use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner.
15. Agrees not to participate in another clinical study during the study period unless the study is in the follow up phase and it has been 1 month since the subject received any experimental agents or treatments. The subject also agrees not to participate in an investigational drug study for at least 1 month after last procedure day.
16. Agrees not to donate blood to a blood bank throughout participation in the study and for at least 2 months after last procedure day.
17. Have a normal ECG; must not have the following to be acceptable: pathologic Q wave abnormalities, significant ST-T wave changes, left ventricular hypertrophy, right bundle branch block, left bundle branch block (sinus rhythm is between 55-100 beats per minute).

Exclusion Criteria:

1. Women who are pregnant or lactating or have a positive serum pregnancy test at enrollment or positive urine pregnancy test on the morning of the first day of any procedure session.
2. Smokers (current use or use over the previous 12 months of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, gum, patch or electronic cigarettes)).
3. Participation in any ongoing investigational drug trial or clinical drug trial period unless the study is in the follow up phase and it has been ≥ 1 month since the subject received any experimental agents or treatments..
4. Abnormal vital signs, defined as:

   * Hypertension (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg) at rest on 2 separate days.
   * Heart rate <55 at rest on 2 separate days
   * Respiratory rate ≤ 11 to ≥ 18 breaths per minute
5. Temperature >38.0ºC (100.4ºF) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 7 days of application of the scopolamine TDDS.
6. History of chronic obstructive pulmonary disease.
7. Positive urine drug screening test.
8. Use of any prescription medication during the period 0 to 30 days or over-the counter medication during the period 0 to 3 days before entry to the study (vitamins, herbal supplements and birth control medications not included).
9. Use of medications or treatments that would significantly influence or exaggerate responses to the test product or that would alter inflammatory or immune response to the product (e.g. antihistamines [within 72 hours prior to dosing], systemic or topical corticosteroids [within 3 weeks prior to dosing], cyclosporine, tacrolimus, cytotoxic drugs, immune globulin, Bacillus Calmette-Guerin [BCG], monoclonal antibodies, radiation therapy).
10. Donation or loss of greater than one pint of blood within 60 days of entry to the study.
11. Any prior serious adverse reaction or hypersensitivity to scopolamine, or any of the inactive ingredients in the TDDS (light mineral oil, polyisobutylene, polypropylene and aluminized polyester film).
12. Have a diagnosis of schizophrenia or other major psychiatric diagnosis.
13. Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month before enrollment in this study or expects to receive an experimental agent during the study.
14. Medical history of a serious chronic condition, including (but not limited to): allergic conditions such as anaphylaxis, asthma or generalized drug reactions; any seizure disorder; glaucoma (open or closed angle); history of pyloric or urinary bladder neck obstruction; intestinal obstruction; difficulty swallowing; stomach or bowel problems (e.g, blockage, muscle weakness, ulcerative colitis, Crohn's disease); bleeding disorders; acid reflux disease; myasthenia gravis; allergy to belladonna alkaloids; impaired hepatic or renal function.
15. Any condition that would, in the opinion of the MAI, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
16. Inability to communicate or co-operate with the investigators.
17. Medical history of significant dermatologic diseases or conditions, such as atopy, psoriasis, vitiligo or conditions known to alter skin appearance or physiologic response (e.g. diabetes, porphyria).
18. History of significant dermatologic cancers (e.g. melanoma, squamous cell carcinoma), except basal cell carcinomas that were superficial and did not involve the investigative site.
19. History of consumption of alcohol within 24 hours prior to dose administration.
20. Subject has an obvious difference in skin color between arms or the presence of a skin condition, excessive hair at the application site, sunburn, raised moles and scars, open sores at application site, scar tissue, tattoo, or coloration that would interfere with placement of test articles, skin assessment, or reactions to drug.
21. Use of monoamine oxidase inhibitors 21 days prior to study.
22. Within 4 weeks prior to dosing, use of medications or treatments that would significantly influence or exaggerate responses to the test product or that would alter inflammatory or immune response to the product or agents deemed to be immunosuppressive as determined by physician investigator.
23. Planned MRI scan of the head during TDDS wear.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at the University of Iowa by advertisements in the "Noon News", a UIHC newsletter, and by a mass email that was sent to all staff/faculty/and students. Recruitment began in November 2016 and continued until the enrollment goal of 24 participants completing all arms of the study was reached in March 2017.
Groups:
- Transderm Scop®, Then IV Scopolamine Hydrbromide: Participants wore a Transderm Scop® patch (1.5 mg) for 3 days and received a single intravenous dose of 0.4 mg scopolamine hydrobromide in a crossover design with adequate washout in between.
- IV Scopolamine HBr, Then Transderm Scop®: Participants received a single intravenous dose of 0.4 mg scopolamine hydrobromide and will wore a Transderm Scop® patch (1.5 mg) for 3 days in a crossover design with adequate washout in between.
Period: First Intervention (3 - 6 Days)
Arm/Group | Transderm Scop®, Then IV Scopolamine Hydrbromide | IV Scopolamine HBr, Then Transderm Scop®
Started | 14 (More subjects not enrolled after consent in other group leaving uneven number.) | 12
Completed | 14 | 12
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Transderm Scop®, Then IV Scopolamine Hydrbromide | IV Scopolamine HBr, Then Transderm Scop®
Started | 14 | 12
Completed | 13 | 10
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 0 | 1
Period: 2nd Intervention (3 - 6 Days)
Arm/Group | Transderm Scop®, Then IV Scopolamine Hydrbromide | IV Scopolamine HBr, Then Transderm Scop®
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis of all study participants that received both the Transderm Scop® (1.5mg/72 hrs) patch and the intravenous scopolamine hydrobromide (0.4mg) injection
Groups:
- All Study Participants: Each of the subjects received Transderm Scop® (1.5mg/72 hrs) and intravenous scopolamine hydrobromide (0.4 mg)
Arm/Group | All Study Participants
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.32 (6.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 21
  African American/Black | 2
  Asian | 1
  Bi-/Multiracial | 1
  Other/Chose not to answer | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.3 (2.88)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Maximum Serum Concentration of Scopolamine (Cmax)
Time Frame: Measured at time points: pre-dose, 1,2,3,4,5,6,8,10,12,24,36,48,60, and 72 hours during Intervention: Transderm Scop® and at time points: pre-dose, 2.5,5,10,20,30,45 minutes, 1.5,2,3,4,5,6,8,10,12 hours during Intervention: scopolamine HBr
Population: The number of participants analyzed represents the total number of participants that completed both interventions.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Transderm Scop®: All participants that received the Transderm Scop® (1.5mg/72 hrs) regardless of assigned arm
- Intravenous Scopolamine Hydrobromide: All participants that received the intravenous scopolamine hydrobromide injection (0.4 mg) regardless of assigned arm
Arm/Group | Transderm Scop® | Intravenous Scopolamine Hydrobromide
Number analyzed (Participants) | 23 | 23
ng/ml | 0.14 (0.08) | 2.63 (1.02)

2. Secondary Outcome: Assessment of Scopolamine Clearance (CL)
Description: This will be done only after the IV is administered to estimate the rate of removal of scopolamine from the body. Will not be measured during patch arm.
Time Frame: Measured at time points: 2.5,5,10,20,30,45 minutes, 1.5,2,3,4,5,6,8,10,12,24,36,48 hours during Intervention: scopolamine HBr
Measure: Mean (Standard Deviation); unit: L/hr
Groups:
- Intervention: IV Scopolamine Hydrobromide: Each of the subjects will receive a single intravenous dose of 0.4 mg scopolamine hydrobromide
  Intravenous scopolamine hydrobromide: 0.4 mg via intravenous injection
Arm/Group | Intervention: IV Scopolamine Hydrobromide
Number analyzed (Participants) | 23
L/hr | 164.4 (48.8)

3. Secondary Outcome: Measurement of Volume of Scopolamine Distribution (V)
Description: This measure is only analyzed for the IV scopolamine HBr arm of the study.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: L
Groups:
- Intravenous Scopolamine Hydrobromide: Each of the subjects will receive a single intravenous dose of 0.4 mg scopolamine hydrobromide
Arm/Group | Intravenous Scopolamine Hydrobromide
Number analyzed (Participants) | 23
L | 488.3 (191.2)

4. Secondary Outcome: Measurement of Elimination Rate Constant of Scopolamine (Kel)
Time Frame: Measured at time points: 73,74,78,84,96,108,120 hours during Intervention: Transderm Scop® and at time points: pre-dose, 2.5,5,10,20,30,45 minutes, 1.5,2,3,4,5,6,8,10,12 hours during Intervention: scopolamine HBr
Measure: Mean (Standard Deviation); unit: 1/hr
Groups:
- Transderm Scop®: Each of the subjects will wear the Transderm Scop® patch (1.5 mg) for 3 days
  Transderm Scop®: TDDS dosage is 1.5 mg/72 hrs
Arm/Group | Transderm Scop® | Intravenous Scopolamine Hydrobromide
Number analyzed (Participants) | 23 | 23
1/hr | 0.06 (0.02) | 0.23 (0.12)

5. Secondary Outcome: Measurement of Time of Maximum Serum Scopolamine Concentration (Tmax)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Transderm Scop® | Intravenous Scopolamine Hydrobromide
Number analyzed (Participants) | 23 | 23
hr | 9.65 (2.21) | 0.04 (0.03)

6. Secondary Outcome: Determination of Area Under the Serum Concentration-time Curve (AUC)
Time Frame: Measured at time points:1,2,3,4,5,6,8,10,12,24,36,48,60,72,73,74,78,84,96,108,120 hours during Intervention: Transderm Scop® and at time points: 2.5,5,10,20,30,45 minutes, 1.5,2,3,4,5,6,8,10,12,24,36, and 48 hours during Intervention: scopolamine HBr
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Transderm Scop® | Intravenous Scopolamine Hydrobromide
Number analyzed (Participants) | 23 | 23
ng*hr/ml | 8.01 (2.8) | 2.6 (0.7)

7. Secondary Outcome: Residual Drug Analysis in Worn TDDS
Description: This will be done in the TDDS after its removal to estimate total amount of absorbed scopolamine.
Time Frame: 3 - 6 months
Measure: Mean (Standard Deviation); unit: % residual drug recovery
Arm/Group | Transderm Scop®
Number analyzed (Participants) | 24
% residual drug recovery | 34.4 (7.7)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected in real time as subjects participated in the study. The study was completed in 5 months.
Groups:
- Intervention: Transderm Scop® (6 Days): Transderm Scop® patch (1.5 mg) for 3 days with 3 days of follow up sample collection time points
  Transderm Scop®: TDDS dosage is 1.5 mg/72 hrs
- Intervention: Intravenous Scopolamine Hydrobromide (3 Days): 0.4 mg of intravenous scopolamine hydrobromide
  Intravenous scopolamine hydrobromide: 0.4 mg via intravenous injection
Arm/Group | Intervention: Transderm Scop® (6 Days) | Intervention: Intravenous Scopolamine Hydrobromide (3 Days)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 24/24 | 25/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: Transderm Scop® (6 Days) (N=24) | Intervention: Intravenous Scopolamine Hydrobromide (3 Days) (N=25)
Decreased Blood Pressure (General disorders) | 10 (15) | 13 (37)
Increased Blood Pressure (General disorders) | 4 (7) | 6 (8)
Decreased Heart Rate (General disorders) | 11 (63) | 15 (73)
Increased Heart Rate (General disorders) | 1 (5) | 2 (3)
Dry Mouth (General disorders) | 14 (31) | 4 (10)
Headache (General disorders) | 2 (2) | 3 (7)
Dilated Pupils (General disorders) | 2 (2) | 6 (6)
Nausea (General disorders) | 2 (2) | 4 (10)
Emesis (General disorders) | 0 (0) | 3 (3)
Dizziness (General disorders) | 3 (5) | 18 (62)
Blurry Vision (General disorders) | 8 (36) | 3 (7)
Fatigue (General disorders) | 5 (9) | 14 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT03029650/Prot_SAP_000.pdf